CLINICAL TRIAL: NCT01290835
Title: Conformal Partial Breast Irradiation With CyberKnife After Resection for Early Stage Breast Cancer
Acronym: CKPBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Essentia Health (Other)
Responsible Party: Principal Investigator, Ken Dornfeld, Radiation Oncologist, Essentia Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMDC10101
Record Dates: First submitted 2011-02-04; First posted 2011-02-07 (Estimated); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: Stereotactic radiotherapy; CyberKnife following lumpectomy; Breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stereotactic radiotherapy (Experimental): Accelerated stereotactic radiotherapy as an adjuvant treatment for early stage breast cancer.
  Interventions: Radiation: Stereotactic radiotherapy delivered by CyberKnife; Radiation: stereotactic radiotherapy

INTERVENTIONS:
Radiation: Stereotactic radiotherapy delivered by CyberKnife — Adjuvant radiotherapy will be delivered using CyberKnife radiotherapy using twice daily sessions for five days for a total of ten sessions.
  Other Names: CyberKnife
Radiation: stereotactic radiotherapy

SUMMARY:
The purpose of this study is to determine if it is feasible, safe, and effective to use Cyberknife radiotherapy to deliver partial breast radiotherapy after lumpectomy.Patients meeting eligibility criteria will be invited to participate. Adjuvant radiotherapy will be delivered using CyberKnife radiotherapy using twice daily sessions for five days for a total of ten sessions. Short-term and long-term toxicity will be assessed as well as Tumor control and site of failure (if any).

DETAILED DESCRIPTION:
This study will determine the feasibility and toxicity of a short course of accelerated radiotherapy as adjuvant treatment for early stage breast cancer. Successful completion of this project may provide a rationale to offer this treatment for select patients with the benefit of potentially less tissue damage and a shorter overall course of therapy. These improvements may ultimately allow more patients the opportunity of breast conserving therapy to treat their cancer

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of breast malignancy, stage T1
2. Surgical treatment with lumpectomy
3. age 60 or older
4. resection margins negative by at least 2mm
5. any grade
6. ER positive
7. unicentric
8. invasive ductal
9. pathologic free of nodal metastases (N0, i- or i+)
10. Post-lumpectomy cavity to whole breast ratio must be less than or equal to 30%

Exclusion criteria

1. Prior radiotherapy to the breast
2. Neoadjuvant chemotherapy
3. multicentric disease
4. Pure DCIS histology
5. Presence of extensive intraductal component
6. Node positive disease (N1 or greater)

Ages: 60 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-06; Primary Completion 2025-08 (Actual); Study Completion 2025-08 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility of using CyberKnife radiotherapy to deliver partial breast radiotherapy for early stage breast cancer. | one year
  Subjects will undergo a treatment plan for partial breast irradiation with cyberknife. Feasibility will be determined by monitoring the number of potential eligible subjects enrolled that can be treated while also respecting normal tissue tolerances.

SECONDARY OUTCOMES:
To determine if conformal irradiation to the operative bed using CyberKnife produces acceptable local control | 1 year
  Subjects will be followed for disease control following standard guidelines that include periodic PE and imaging with either mammography or screening breast MRaI for 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Ken Dornfeld, MD, Principal Investigator — Essentia Health Oncology
Locations (1):
- Essentia Health SMDC Cancer Center, Duluth, Minnesota, United States

REFERENCES:
- [Background] Fisher B, Jeong JH, Anderson S, Bryant J, Fisher ER, Wolmark N. Twenty-five-year follow-up of a randomized trial comparing radical mastectomy, total mastectomy, and total mastectomy followed by irradiation. N Engl J Med. 2002 Aug 22;347(8):567-75. doi: 10.1056/NEJMoa020128. PMID 12192016
- [Background] Fisher B, Anderson S, Bryant J, Margolese RG, Deutsch M, Fisher ER, Jeong JH, Wolmark N. Twenty-year follow-up of a randomized trial comparing total mastectomy, lumpectomy, and lumpectomy plus irradiation for the treatment of invasive breast cancer. N Engl J Med. 2002 Oct 17;347(16):1233-41. doi: 10.1056/NEJMoa022152. PMID 12393820
- [Background] Clarke M, Collins R, Darby S, Davies C, Elphinstone P, Evans V, Godwin J, Gray R, Hicks C, James S, MacKinnon E, McGale P, McHugh T, Peto R, Taylor C, Wang Y; Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Effects of radiotherapy and of differences in the extent of surgery for early breast cancer on local recurrence and 15-year survival: an overview of the randomised trials. Lancet. 2005 Dec 17;366(9503):2087-106. doi: 10.1016/S0140-6736(05)67887-7. PMID 16360786
- [Background] Holland R, Veling SH, Mravunac M, Hendriks JH. Histologic multifocality of Tis, T1-2 breast carcinomas. Implications for clinical trials of breast-conserving surgery. Cancer. 1985 Sep 1;56(5):979-90. doi: 10.1002/1097-0142(19850901)56:53.0.co;2-n. PMID 2990668
- [Background] Veronesi U, Marubini E, Mariani L, Galimberti V, Luini A, Veronesi P, Salvadori B, Zucali R. Radiotherapy after breast-conserving surgery in small breast carcinoma: long-term results of a randomized trial. Ann Oncol. 2001 Jul;12(7):997-1003. doi: 10.1023/a:1011136326943. PMID 11521809
- [Background] Clark RM, Whelan T, Levine M, Roberts R, Willan A, McCulloch P, Lipa M, Wilkinson RH, Mahoney LJ. Randomized clinical trial of breast irradiation following lumpectomy and axillary dissection for node-negative breast cancer: an update. Ontario Clinical Oncology Group. J Natl Cancer Inst. 1996 Nov 20;88(22):1659-64. doi: 10.1093/jnci/88.22.1659. PMID 8931610
- [Background] Holli K, Saaristo R, Isola J, Joensuu H, Hakama M. Lumpectomy with or without postoperative radiotherapy for breast cancer with favourable prognostic features: results of a randomized study. Br J Cancer. 2001 Jan;84(2):164-9. doi: 10.1054/bjoc.2000.1571. PMID 11161371
- [Background] Liljegren G, Holmberg L, Bergh J, Lindgren A, Tabar L, Nordgren H, Adami HO. 10-Year results after sector resection with or without postoperative radiotherapy for stage I breast cancer: a randomized trial. J Clin Oncol. 1999 Aug;17(8):2326-33. doi: 10.1200/JCO.1999.17.8.2326. PMID 10561294
- [Background] Schroen AT, Brenin DR, Kelly MD, Knaus WA, Slingluff CL Jr. Impact of patient distance to radiation therapy on mastectomy use in early-stage breast cancer patients. J Clin Oncol. 2005 Oct 1;23(28):7074-80. doi: 10.1200/JCO.2005.06.032. PMID 16192590
- [Background] Benitez PR, Chen PY, Vicini FA, Wallace M, Kestin L, Edmundson G, Gustafson G, Martinez A. Partial breast irradiation in breast conserving therapy by way of intersitial brachytherapy. Am J Surg. 2004 Oct;188(4):355-64. doi: 10.1016/j.amjsurg.2004.06.027. PMID 15474426
- [Background] Chen PY, Vicini FA, Benitez P, Kestin LL, Wallace M, Mitchell C, Pettinga J, Martinez AA. Long-term cosmetic results and toxicity after accelerated partial-breast irradiation: a method of radiation delivery by interstitial brachytherapy for the treatment of early-stage breast carcinoma. Cancer. 2006 Mar 1;106(5):991-9. doi: 10.1002/cncr.21681. PMID 16421922
- [Background] Benitez PR, Keisch ME, Vicini F, Stolier A, Scroggins T, Walker A, White J, Hedberg P, Hebert M, Arthur D, Zannis V, Quiet C, Streeter O, Silverstein M. Five-year results: the initial clinical trial of MammoSite balloon brachytherapy for partial breast irradiation in early-stage breast cancer. Am J Surg. 2007 Oct;194(4):456-62. doi: 10.1016/j.amjsurg.2007.06.010. PMID 17826055
- [Background] Vicini F, Winter K, Wong J, Pass H, Rabinovitch R, Chafe S, Arthur D, Petersen I, White J, McCormick B. Initial efficacy results of RTOG 0319: three-dimensional conformal radiation therapy (3D-CRT) confined to the region of the lumpectomy cavity for stage I/ II breast carcinoma. Int J Radiat Oncol Biol Phys. 2010 Jul 15;77(4):1120-7. doi: 10.1016/j.ijrobp.2009.06.067. Epub 2009 Nov 10. PMID 19910132
- [Background] Hepel JT, Tokita M, MacAusland SG, Evans SB, Hiatt JR, Price LL, DiPetrillo T, Wazer DE. Toxicity of three-dimensional conformal radiotherapy for accelerated partial breast irradiation. Int J Radiat Oncol Biol Phys. 2009 Dec 1;75(5):1290-6. doi: 10.1016/j.ijrobp.2009.01.009. Epub 2009 Apr 22. PMID 19395195
- [Background] Dornfeld K, Gessert CE, Renier CM, McNaney DD, Urias RE, Knowles DM, Beauduy JL, Widell SL, McDonald BL. Differences in breast tissue oxygenation following radiotherapy. Radiother Oncol. 2011 Aug;100(2):289-92. doi: 10.1016/j.radonc.2011.02.004. Epub 2011 Feb 26. PMID 21356563
- [Background] Smith BD, Arthur DW, Buchholz TA, Haffty BG, Hahn CA, Hardenbergh PH, Julian TB, Marks LB, Todor DA, Vicini FA, Whelan TJ, White J, Wo JY, Harris JR. Accelerated partial breast irradiation consensus statement from the American Society for Radiation Oncology (ASTRO). Int J Radiat Oncol Biol Phys. 2009 Jul 15;74(4):987-1001. doi: 10.1016/j.ijrobp.2009.02.031. PMID 19545784
- [Background] Le QT, Loo BW, Ho A, Cotrutz C, Koong AC, Wakelee H, Kee ST, Constantinescu D, Whyte RI, Donington J. Results of a phase I dose-escalation study using single-fraction stereotactic radiotherapy for lung tumors. J Thorac Oncol. 2006 Oct;1(8):802-9. PMID 17409963
- [Background] Rose MA, Olivotto I, Cady B, Koufman C, Osteen R, Silver B, Recht A, Harris JR. Conservative surgery and radiation therapy for early breast cancer. Long-term cosmetic results. Arch Surg. 1989 Feb;124(2):153-7. doi: 10.1001/archsurg.1989.01410020023002. PMID 2916935
- [Background] Lovey K, Fodor J, Major T, Szabo E, Orosz Z, Sulyok Z, Janvary L, Frohlich G, Kasler M, Polgar C. Fat necrosis after partial-breast irradiation with brachytherapy or electron irradiation versus standard whole-breast radiotherapy--4-year results of a randomized trial. Int J Radiat Oncol Biol Phys. 2007 Nov 1;69(3):724-31. doi: 10.1016/j.ijrobp.2007.03.055. Epub 2007 May 24. PMID 17524571
- [Background] NCCN Clinical Practice Guidelines in Oncology, V.I.2010,